CLINICAL TRIAL: NCT06276660
Title: Comparing Symptom Provocation and Physiological Response Between Buffalo Concussion Treadmill Test (BCTT) Protocol and Modified Dynamic Exertion Test (mEXiT) Post Concussion
Brief Title: Post-Concussion Differences Between Buffalo Concussion Treadmill Test (BCTT) and Modified Dynamic Exertion (mEXiT) Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Professor, Research Director University of Pittsburgh Concussion Lab, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY23070079
Record Dates: First submitted 2024-02-06; First posted 2024-02-26 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mtbi; concussion; exertion therapy
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buffalo Concussion Treadmill Test (BCTT) (Active Comparator): Participants in this group will complete the Buffalo Concussion Treadmill Test (BCTT). This involves individuals walking at 5.8 km/hr. (3.6 mph) at a 0.0% incline (5.1 km/hr. [3.2 mph] if below 5' 10" tall), the treadmill incline is increased 1 degree each minute for the first 15 minutes, then speed increased 0.64 km/hr. (0.4 mph) each minute thereafter.
  Interventions: Other: BCTT
- Modified EXiT Test (mEXiT) (Experimental): Participants in this group will complete the modified EXiT test (mEXiT). Participants will complete a 12 minute treadmill interval program followed by a dynamic circuit (10 squat jumps, 10 side to side push ups and 10 medicine ball rotations), jump ball toss, zig zag agility and arrow agility. Parameters will be recorded the same as the established dynamic EXiT test; heart rate and RPE will be recorded at 0, 2, 6:30 and 12 minutes of the treadmill program as well as after the second trial of each activity. The time to complete two trials of the zig zag agility and arrow agility will also be recorded.
  Interventions: Other: Dynamic ExIT

INTERVENTIONS:
Other: BCTT — Participants will complete the Buffalo Concussion Treadmill Test, which involves individuals walking at 5.8 km/hr. (3.6 mph) at a 0.0% incline (5.1 km/hr. [3.2 mph] if below 5' 10" tall), the treadmill incline is increased 1 degree each minute for the first 15 minutes, then speed increased 0.64 km/hr. (0.4 mph) each minute thereafter.
  Arms: Buffalo Concussion Treadmill Test (BCTT)
Other: Dynamic ExIT — The modified EXiT test will complete a 12 minute treadmill interval program followed by a dynamic circuit (10 squat jumps, 10 side to side push ups and 10 medicine ball rotations), jump ball toss, zig zag agility and arrow agility. Parameters will be recorded the same as the established dynamic EXiT test; heart rate and RPE will be recorded at 0, 2, 6:30 and 12 minutes of the treadmill program as well as after the second trial of each activity. The time to complete two trials of the zig zag agility and arrow agility will also be recorded.
  Arms: Modified EXiT Test (mEXiT)

SUMMARY:
This study aims to compare symptom provocation, physiologic response, and rate of perceived (RPE) between the Buffalo Concussion Treadmill Test (BCTT) and a Modified Dynamic Exertion (mEXiT) test after sport related concussion in adolescents aged 14-17. Participants will be enrolled at their initial concussion clinical visit within 14 days of their injury, and randomly assigned to either the BCTT or mEXiT group. Participants will complete a single visit.

DETAILED DESCRIPTION:
The Buffalo Concussion Treadmill Test is a well established test to determine intensity of exercise without significant symptoms provocation after sport related concussion.

This study will help determine if there is a difference in type of symptom response between the two tests, due to the dynamic changes of direction and strain on the vestibular system with the m-EXiT group. The investigators hypothesize there will not be a significant difference between the two groups in time to clearance to return to sport despite allowing for higher symptoms earlier on in recovery.

High school athletes who have been diagnosed with a sport-related concussion will be randomly assigned to complete either the BCTT or the modified dynamic EXiT test (m-EXiT). The BCTT group will follow the established protocol and exercise to an increase of 2/10 symptoms on a visual analog scale (VAS) or 17/20 on rate of perceived effort (RPE) scale. The m-EXiT test will complete a shortened version of the dynamic EXiT test, but will stop if participants have an increase of greater than 4 points of headache, dizziness or nausea or RPE of 17/20. Symptoms, heart rate, and RPE will be measured through out both tests as well as Post-Concussion Symptom Scale (PCSS), Vestibular Ocular Motors Screening (VOMS), blood pressure and heart rate will be administered before and after testing. The time (in days) to recovery, will also be recorded from the medical record to determine if there is a difference between the two groups.

The primary outcome for the study will be symptoms post test and heart rate. Secondary measures include: Post Concussion Symptom Score (PCSS), Clinical Profiles Screening (CP-Screen), Vestibular Ocular Motor Screening (VOMS), Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder - 7 (GAD-7) and blood pressure. These will be collected at one visit with participants, there are no follow-up or subsequent visits for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a sport related concussion within 14 days of injury
* Participants referred to exertion therapy after a trained clinician from University of Pittsburgh Medical Center (UPMC) Sports Medicine Concussion Program has interpreted neurocognitive, vestibular, and clinical interview outcomes and determined the participant is capable of completing structured exercise.

Exclusion Criteria:

* Medically cleared from a previous concussion within the past 6 months
* More than 2 previous concussions (excluding current injury)
* History of brain surgery or traumatic brain injury (TBI) (based on Glasgow Coma Scale of <13)
* History of neurological disorder (seizure disorder, epilepsy, brain tumors or malformations)
* Current history of pre-existing vestibular disorder or oculomotor condition
* Currently taking antidepressant, anticoagulant, beta-blocker, or anticonvulsant prescription medications
* Incapable of treadmill running up to 5.5 miles per hour (mph) and 4.5 mph for males and females respectively (self-reported).
* Diagnosed with a cardiac, peripheral, or cerebrovascular disease (type 1 or 2 diabetes, or renal disease.
* Experienced chest pain or shortness of breath while at rest or with mild exertion.
* Lose balance because of dizziness or have lost consciousness (aside from concussion) from exertion
* Currently have (or have had within the past 12 months) a bone, joint, or soft tissue (muscle, ligament, or tendon) problem that could be made worse by physical activity
* Been told by a doctor to only conduct physical activity under medical supervision.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Physiological response to dynamic or aerobic test (HEART RATE) | Visit 1 (baseline) (pre, during, and post testing) 90 minutes
  Participants will have their heart rate taken before the exercise protocol, then monitored throughout the test and after they complete the BCTT or mEXiT.
Physiological response to dynamic or aerobic test (SYMPTOM PROVOCATION) | Visit 1 (baseline) (pre and post testing) 90 minutes
  Participants will report on a Likert scale ranging from 0-10 (10 being severe) for headache, dizziness, and nausea, and provide a rating of perceived exertion (RPE) on a Borg scale ranging from 6 to 20 before and after completion of the BCTT or mEXiT.

SECONDARY OUTCOMES:
Post Concussion Symptom Scale | Visit 1 Baseline (60-90 minutes), participants only complete one visit
  Participants rate on a 7 point Likert scale the presence and severity of 22 common concussion-related symptoms, including, but not limited to headache, dizziness, confusion, fogginess. The scale is 0-6 (0=none, 1-2=mild, 3-4=moderate, 5-6=severe). Higher the score, the more symptoms participant is reporting.
Patient Health Questionnaire (PHQ-9) | Visit 1 Baseline (60-90 minutes), participants only complete one visit
  The PHQ-9 is a 9 item questionnaire that assesses the presence and severity of depression over the last 2-weeks. Total score ranges from 1-27, with higher scores indicating higher level of depression. Scale is 0-4 (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day). Higher scores indicate worse reporting of issues.
Generalized Anxiety Disorder (GAD-7) | Visit 1 Baseline (60-90 minutes), participants only complete one visit
  The GAD-7 is a seven item self-reported questionnaire that measures severity of symptoms regarding anxiety. Responses are 0 = not at all, 1 = several days, 2= more than half the days, and 3 = nearly every day. Higher scores are indicative of higher anxiety (0-4 = minimal anxiety, 5-9= mild anxiety, 10-14 =moderate anxiety, 15-21 = severe anxiety (higher scores indicate higher level of reported anxiety).
Vestibular Ocular Motor Screening (VOMS) | Visit 1 Baseline (pre and post testing 60-90 minutes), participants only complete one visit
  Participants will complete a VOMS assessment which will take approximately 5 minutes. Prior to screening, the participant reports baseline symptoms (headache, dizziness, nausea, fogginess) on a scale from 0 to 10. Then the participant performs different eye movements that include: smooth pursuits, saccades (horizontal & vertical), convergence, vestibular ocular reflex (VOR [horizontal & vertical]), visual motor sensitivity (VMS) and again rates his/her symptoms (headache, dizziness, nausea, fogginess) on a Likert scale from 0 to 10. Abnormal findings or provocation of symptoms with any test may indicate dysfunction. This will be completed by a clinician or researcher. This procedure will be repeated after BCTT and mEXiT protocol on the same day. Higher scores indicate worse symptoms.
Clinical Profiles Screening (CP-Screen) | Visit 1 Baseline (60-90 minutes), participants only complete one visit
  The CP Screen is a 29 item self-report, clinical profiles based symptom inventory that measures five concussion clinical profiles: 1) anxiety/mood, 2) cognitive/fatigue, 3) migraine, 4) ocular, 5) vestibular; and two modifying factors, sleep and cervical. Patients rate the severity of their symptoms as none = 0, mild = 1, moderate = 2, or severe =3. Scores are totaled across the clinical profiles and symptom modifiers. The measure also yields a CP-Screen total raw score ranging from (0-87) with higher scores reflecting more symptoms.
Blood Pressure | Visit 1 Baseline (pre and post testing 60-90 minutes), participants only complete one visit
  Participants blood pressure will be taken same-day, before and after the BCTT or mEXiT test (both systolic and diastolic BP will be recorded with all measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Kontos, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC/Univ of Pgh Sports Medicine Concussion Research Program, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers who sent a request to to the study investigators. The data can be used for any analysis purpose, including publications or presentations.
  After de-identification, all of the individual participant data collected during the trial will be available for sharing.
Supporting Information: Study Protocol
Time Frame: During and after study completion. No end date
Access Criteria: Researchers will need to contact the study investigators and ask for access to available de-identified data.